CLINICAL TRIAL: NCT06198647
Title: Effect of Tui-Na Versus Positional Release Techniques on Pregnancy Related Low Back Pain in the Third Trimester. A Randomized Trial
Brief Title: Manual Therapy for Pregnancy Related Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Aliaa Mohamed Elabd, lecturer, basic science department, faculty of physical therapy, benha university, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT.BU.EC.2
Record Dates: First submitted 2023-12-07; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: manual therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tui-na (Experimental): Application of tui-na techniques for the women while being in prone lying position.
  Interventions: Procedure: Tui-na massage
- positional release techniques (Active Comparator): Application of positional release techniques for the women while being in prone lying position.
  Interventions: Procedure: positional release technique

INTERVENTIONS:
Procedure: Tui-na massage — Using Tui-na massage for the back muscles
  Arms: tui-na
Procedure: positional release technique — using positional release manual technique to relax the back muscles
  Arms: positional release techniques

SUMMARY:
More than 50% of women experience pain in the lumbopelvic area during pregnancy. The prevalence of pain increases with the duration of pregnancy. Trunk muscles are needed to sustain low levels of activity for an extended duration. Preventing muscles from fatiguing is very important. Manual therapy techniques can minimize loading of the spine while improving muscular endurance and preventing fatigue. Moreover, inhibition of the trigger points of the spinal musculature is an important factor to consider.

DETAILED DESCRIPTION:
Tui-Na massage and positional release therapy are both of the common manual therapies used recently for low back pain. However, no studies have compared their effects on pregnancy related low back pain in third trimester.

ELIGIBILITY:
Inclusion Criteria:

* low back pain
* mild to moderate disability concurring to the Oswestry Disability Index (up to 40%),
* age ranged from 20 - 40 years

Exclusion Criteria:

* Current physical therapy or medical treatment for low back pain,
* contracture or surgery affecting the lumbar spine,
* scoliosis,
* pathologies such as inflammatory diseases,
* skin diseases,
* congenital diseases,
* neurological diseases,
* dislocations, neoplasms,
* disc prolapse,
* visual or auditory problems

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant females
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
back pain intensity | through study completion, an average of 2 months
  will be measure by the visual analogue scale that range from 0 to 10 with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
The pressure pain threshold (kg/cm2) | through study completion, an average of 2 months
  will be measured using a pressure algometer that will be placed vertically on the most tender point at the low back para spinal muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa M Elabd, Principal Investigator — Benha University
Locations (1):
- Benha University, Cairo, Benah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: upon completion
Access Criteria: URL will be created after the ending of data acquisition.

REFERENCES:
- [Derived] Elabd AM, Hasan S, Alghadir AH, Elabd OM, Shawky GM, Iqbal A, Marwan YN. Effect of Tui-Na versus positional release techniques on pregnancy-related low back pain in the third-trimester: A randomized comparative trial. Medicine (Baltimore). 2024 Dec 13;103(50):e40879. doi: 10.1097/MD.0000000000040879. PMID 39686497